CLINICAL TRIAL: NCT06406244
Title: Efficacy of Transcutaneous Electrical Acupoint Stimulation on Chronic Pain and Survival in Patients Undergoing Hepatectomy: a Prospective, Randomized Controlled Trial
Brief Title: Efficacy of TEAS on Chronic Pain and Survival in Patients Undergoing Hepatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024HX1564-2
Record Dates: First submitted 2024-05-05; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients who meet the enrollment criteria will be randomized 1:1 to either the transcutaneous electrical acupoint stimulation (TEAS group) or the sham groups using a computer-generated random number table.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of participants will be maintained throughout the observation period. The sham group will receive electrode attachment but without stimulation. Throughout the study, for adequate blinding, an opaque tape will be applied to the patient's skin above the electrodes, and the patient's target acupoints will be wrapped in a blanket. All patients will be informed that they might or might not feel a tingling sensation around the acupoints when the TEAS device is working. The patients should not be unblinded until the statistical analysis of the study data is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS group (Experimental): Patients who meet the enrollment criteria will be randomized 1:1 to either the transcutaneous electrical acupoint stimulation (TEAS）or the sham groups. In the TEAS group, the acupoints are bilateral neiguan (PC6), Hegu (L14), Yanglingquan (GB34), Zusanli (ST 36) and Renying (ST9) acupoints. Patients will receive 30 min TEAS before anesthesia until be discharged from the post-anaesthesia care unit (PACU). The same treatment for 30 min will be performed on the 1st, 2nd and 3rd days after surgery.The stimulation intensity will be adjusted in accordance with the maximal level tolerated by each patient.
  Interventions: Device: TEAS group
- Sham group (Placebo Comparator): Patients in the sham group will receive electrodeattachment but without stimulation.
  Interventions: Device: sham group

INTERVENTIONS:
Device: TEAS group — Transcutaneous electrical acupoint stimulation (TEAS) is a contemporary modification of traditional acupuncture that sends electrical impulses into acupoints through electrodes on the skin surface. In the TEAS group, patients will receive TEAS 30 min before anesthesia until be discharged from the post-anaesthesia care unit (PACU). The same treatment will be performed on the 1st, 2nd and 3rd days after surgery. The stimulation intensity will be adjusted in accordance with the maximal level tolerated by each patient.
  Arms: TEAS group
Device: sham group — Patients in the sham group will receive electrode attachment but without stimulation.
  Arms: Sham group

SUMMARY:
This study is a further observation and follow-up of the patients enrolled in the registration number NCT06341270 to further evaluate the efficacy of TEAS on postoperative chronic pain, quality of life and survival rate in patients undergoing hepatectomy.

DETAILED DESCRIPTION:
This study is a further observation and follow-up of the patients enrolled in the registration number NCT06341270 to further evaluate the efficacy of TEAS on postoperative chronic pain and survival in patients undergoing hepatectomy. Patients who meet the enrollment criteria will be randomized 1:1 to either the transcutaneous electrical acupoint stimulation (TEAS）or the sham groups. In the TEAS group, the acupoints are bilateral neiguan (PC6), Hegu (L14), Yanglingquan (GB34), Zusanli (ST 36) and Renying (ST9) acupoints. Patients will receive TEAS 30 min before anesthesia until being discharged from the post-anaesthesia care unit (PACU). The same treatment for 30 min will be performed on the 1st, 2nd and 3rd days after surgery. The stimulation intensity will be adjusted in accordance with the maximal level tolerated by each patient. Patients in the sham group will receive electrode attachment but without stimulation. Follow-up after discharge includes chronic pain, the impact of chronic pain on quality of life, the relapse-free survival, overall survival at 3 months and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80 years old; ASA physical status classⅠ-Ⅲ; Patients scheduled for elective hepatectomy.

Exclusion Criteria:

Have a history of epilepsy; Rash or local infection over the acupoint stimulation skin area; Pregnancy or breastfeeding; Mental retardation, psychiatric, or neurological disease; Inability to comprehend the numeric rating scale (NRS); Implantation of a cardiac pacemaker, cardioverter, or defibrillator; Chronic opioid use; Metastases in other organs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of chronic pain at 3 months postoperatively | 3 months postoperatively
  Chronic pain is defined as pain that lasts or recurs for longer than 3 months. For chronic postsurgical pain(CPSP), it mainly refers to the pain that persists past normal healing time. Pain scoring is performed at 3 months using the Numerical Rating Scale(NRS), with 11 digits ranging from 0 to 10 indicating the degree of pain, 0 indicating no pain, and 10 indicating severe pain. Subjects choose a number to indicate the degree of pain based on their personal pain experience.

SECONDARY OUTCOMES:
The incidence of chronic pain at 6 months | 6 months postoperatively
  Chronic pain is defined as pain that lasts or recurs for longer than 3 months. For chronic postsurgical pain(CPSP), it mainly refers to the pain that persists past normal healing time. Pain scoring is performed at 3 months using the Numerical Rating. Scale(NRS), with 11 digits ranging from 0 to 10 indicating the degree of pain, 0 indicating no pain, and 10 indicating severe pain. Subjects choose a number to indicate the degree of pain based on their personal pain experience.
Overall survival postoperatively | Up to 6 months postoperatively
  Overall survival is defined as the time between the date from surgery to the date of death.
Recurrence-free survival postoperatively | Up to 6 months postoperatively
  Postoperative re-examination is based on the diagnosis of enhanced CT, MRI, ultrasound or blood examination todetermine whether the patient has recurrence and metastasis. Recurrence-free time refers to the time from surgery to tumor recurrence based on the above CT, MRI, etc.
Disability-free survival postoperatively | Up to 6 months postoperatively
  Patient self-assessment is carried out by using the World Health Organization(WHO) Disability Scale, with a minimum score of 12 points and a maximum score of 60 points. The lower the score, the higher the quality of life.
Quality of Recovery Scale Score postoperatively | Up to 6 months postoperatively
  The global QoR-15 score ranges from 0 to 150 and is categorized as five quality of recovery dimensions, including physical comfort(5 items), emotional state(4 items), psychological support(2 items), physical independence(2 items), and pain(2 items). Each piece is graded using an 11-point Likert scale. The QoR is classified according to the QoR-15 score as excellent(QoR-15 > 135), good(122 ≤ QoR-15 ≤ 135), moderate(90 ≤ QoR-15 ≤ 121) and poor(QoR-15 <90).
The sleep quality score postoperatively | Up to 6 months postoperatively
  Postoperative sleep quality is evaluated using the Athens Insomnia Scale(AIS). The AIS consists of 8 items: waking up at night, sleep induction, final awakening, total sleep duration, sleep quality, well-being, functional ability, and daytime sleepiness. The AIS score ranges from 0 to 24 points, and a total score of 6 points or higher indicates adiagnosis of insomnia.
The anxiety and depression scores postoperatively | Up to 6 months postoperatively
  Anxiety and depression score will be evaluated using the Hospital Anxiety and Depression Scale(HADS).The HADS consists of 14 questions, with 7 items each for the anxiety and depression subscales. The score for each item ranges from 0 to 3 points, and scores are summed to yield a separate score for anxiety(HADS-A) and depression(HADS-D).
The prevalence of neuropathic pain | Up to 6 months postoperatively
  The ID Pain scale is used as a validated assessment of neuropathic pain. ID pain questionnaire consists of six items. Pain higher scores suggest a neuropathic component to the pain.
Brief Pain Inventory(BPI) pain interference subscale score | Up to 6 months postoperatively
  BPI pain interference subscale is a 7-item questionnaire asking participants to describe how pain has interfered general activity, mood, walking, normal work, relations with others, sleep, and enjoyment of life. Each question is answered on a scale 0(does not interfere) to 10(completely interferes). The total range of score is 0-70. The higher the scores suggest the worse the interference.

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: No